CLINICAL TRIAL: NCT04787471
Title: Randomized Comparison of Standard vs. Accelerated Corneal Crosslinking for Treatment of Corneal Neovascularization With or Without Concomitant Inflammation and/or Infection
Brief Title: Corneal Crosslinking for Treatment of Corneal Neovascularization
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Price Vision Group (Industry)
Collaborators: Cornea Research Foundation of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-001
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Corneal Neovascularization
MeSH Terms: conditions — Corneal Neovascularization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 30 minute photoactivation (Active Comparator): photoactivation of riboflavin 0.1% using 365-nm UV light, 3mW/cm2 for 30 minutes
  Interventions: Combination Product: 30 minute photoactivation of riboflavin 0.1%
- 10 minute photoactivation (Active Comparator): photoactivation of riboflavin 0.1% using 365-nm UV light, 9mW/cm2 for 10 minutes
  Interventions: Combination Product: 10 minute photoactivation of riboflavin 0.1%

INTERVENTIONS:
Combination Product: 30 minute photoactivation of riboflavin 0.1% — Use of riboflavin 0.1% eye drops and 3mW/cm2 UVA light for 30 minutes
  Arms: 30 minute photoactivation
Combination Product: 10 minute photoactivation of riboflavin 0.1% — Use of riboflavin 0.1% eye drops and 9mW/cm2 UVA light for 10 minutes
  Arms: 10 minute photoactivation

SUMMARY:
The study objective is to assess safety and efficacy of photo-activation of riboflavin for treatment of corneal neovascularization with or without concomitant inflammation and/or infection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* With active inflammation or infection causing vascularization and possibly melting of the cornea, or vessels extending into the cornea causing lipid deposition, or vascularization that could significantly increase the risk of rejection of a current or planned corneal transplant, or vessels that continue to extend into the cornea despite topical treatment with corticosteroids.
* Signed written informed consent.

Exclusion Criteria:

* Known sensitivity to treatment medications
* Current condition that in the investigator's opinion could compromise safety or data integrity.
* Pregnancy (including plan to become pregnant) or lactation during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
corneal neovascularization as a proportion of the total corneal area | 6 months
  the cornea will be photographed and morphometric image analysis software will be used to measure corneal neovascularization as a proportion of the total corneal area. The proportion measured at baseline will be compared with the proportion measured at 6 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, Jr., MD, Principal Investigator — Price Vision Group
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hersh PS, Stulting RD, Muller D, Durrie DS, Rajpal RK; U.S. Crosslinking Study Group. U.S. Multicenter Clinical Trial of Corneal Collagen Crosslinking for Treatment of Corneal Ectasia after Refractive Surgery. Ophthalmology. 2017 Oct;124(10):1475-1484. doi: 10.1016/j.ophtha.2017.05.036. Epub 2017 Jun 24. PMID 28655538
- [Background] Hersh PS, Stulting RD, Muller D, Durrie DS, Rajpal RK; United States Crosslinking Study Group. United States Multicenter Clinical Trial of Corneal Collagen Crosslinking for Keratoconus Treatment. Ophthalmology. 2017 Sep;124(9):1259-1270. doi: 10.1016/j.ophtha.2017.03.052. Epub 2017 May 7. PMID 28495149
- [Background] Price MO, Fairchild K, Feng MT, Price FW Jr. Prospective Randomized Trial of Corneal Cross-linking Riboflavin Dosing Frequencies for Treatment of Keratoconus and Corneal Ectasia. Ophthalmology. 2018 Apr;125(4):505-511. doi: 10.1016/j.ophtha.2017.10.034. Epub 2017 Dec 2. PMID 29203068
- [Background] Price MO, Tenkman LR, Schrier A, Fairchild KM, Trokel SL, Price FW Jr. Photoactivated riboflavin treatment of infectious keratitis using collagen cross-linking technology. J Refract Surg. 2012 Oct;28(10):706-13. doi: 10.3928/1081597X-20120921-06. PMID 23062001
- [Background] Schaub F, Hou Y, Zhang W, Bock F, Hos D, Cursiefen C. Corneal Crosslinking to Regress Pathologic Corneal Neovascularization Before High-Risk Keratoplasty. Cornea. 2021 Feb 1;40(2):147-155. doi: 10.1097/ICO.0000000000002406. PMID 33395116
- [Derived] Price FW Jr, Tefasse Z, Frances KD, Feng MT, Gang A, Price MO. Assessment of Corneal Crosslinking for the Treatment of Corneal Neovascularization With and Without Associated Infection. Cornea. 2025 Apr 2. doi: 10.1097/ICO.0000000000003869. Online ahead of print. PMID 40172865